CLINICAL TRIAL: NCT04107701
Title: Indoor Air Quality and Respiratory Morbidity in School-Aged Children With BPD
Acronym: AeroBPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Jonathan M. Gaffin, Principal Investigator, Assistant Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: P00029918; R01ES030100 (NIH)
Record Dates: First submitted 2019-09-24; First posted 2019-09-27 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Bronchopulmonary Dysplasia; Chronic Lung Disease of Newborn; Environmental Exposure
Keywords: BPD; bronchopulmonary dysplasia; children and environment; environment; bronchopulmonary dysplasia and environment; environment and children; chronic lung disease of newborn; environment and chronic lung disease of the newborn
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigators want to learn the role of indoor environmental exposures on respiratory symptoms, and, separately, on lung function deficits in school-aged children with bronchopulmonary dysplasia (BPD).

DETAILED DESCRIPTION:
Bronchopulmonary dysplasia (BPD) is the most common respiratory disease affecting children born prematurely and leads to long-term respiratory symptoms and lung function impairment throughout childhood. This study will, evaluate the contribution of indoor sources of respiratory irritants to respiratory health impairment in school-aged children with BPD. State-of-the-art measures of indoor air quality constituents will assess the relationship of nitrogen dioxide (NO2), particulate matter (PM2.5), as well as, concentrations of allergens (mold, mouse, cockroach, pet), endotoxin, air temperature and humidity with concurrently measured respiratory symptoms and lung function in a well-characterized cohort of children with BPD. This research will identify specific harmful components of the indoor environment associated with respiratory morbidity and poor lung function in children with BPD.

Investigators will ask the participants to come in for a one time clinic visit for undergoing procedures as well as answering questions regarding health and home environment. During the 1 year of participation there will also be 2 home assessment visits where investigators will take a sample of the home environment as well record home characteristics.

ELIGIBILITY:
Inclusion Criteria:

* children 6-12 yrs old
* born <32 wks gestational age
* diagnosis of BPD or > 28 days of oxygen or respiratory support

Exclusion Criteria:

* major airway or chest surgery
* physical or mental impairment that will prevent from doing spirometry
* plans to move out of state within the next 9 months

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 6-12 years with BPD in MA
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory Morbidity | 2 weeks
  maximum symptom days in the prior 2 weeks assessed at completion of home sampling visits ( Units: days scale: 0-14 days with symptoms, higher is worse
Lung Function | 1 yr
  Spirometry (FEV1 percent predicted) Units: percent Scale: continuous integers, higher is better

SECONDARY OUTCOMES:
Lung function | 1 year
  Oscillometry (R5-20)
Lung function | 1 year
  Oscillometry (AX) units: cmH20 scale 0 - infinity, lower is better
Lung function | 1 year
  Oscillometry R5 units: cmH20 scale 0 - infinity, lower is better
Lung function | 1 year
  Oscillometry R5-20 units: cmH20 scale 0 - infinity, lower is better
Lung function | 1 year
  Oscillometry X5 units: cmH20 scale 0 - infinity, lower is better
Lung function | 1 year
  Oscillometry Fres units: Hz scale 0 - infinity, lower is better
Lung Function | 1 year
  FEV1/FVC units: percent scale: continuous integer, higher is better
Lung Function | 1 year
  FVC percent predicted units: percent scale: continuous integer, higher is better
Lung Function | 1 year
  FEF25-75 percent predicted units: percent scale: continuous integer, higher is better

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Gaffin, MD. MMSc., Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Childrens Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruran HB, Adamkiewicz G, Cunningham A, Petty CR, Greco KF, Gunnlaugsson S, Stamatiadis N, Sierra G, Vallarino J, Alvarez M, Hayden LP, Sheils CA, Weller E, Phipatanakul W, Gaffin JM. Air quality, Environment and Respiratory Outcomes in Bronchopulmonary Dysplasia, the AERO-BPD cohort study: design and adaptation during the SARS-CoV-2 pandemic. BMJ Open Respir Res. 2021 Jun;8(1):e000915. doi: 10.1136/bmjresp-2021-000915. PMID 34193433